CLINICAL TRIAL: NCT01881815
Title: Swab Sample Collection for the Detection of Bacterial Proteases in Wounds Assay
Brief Title: Swab Sample Collection for the Detection of Bacterial Proteases
Status: Completed | Type: Observational
Sponsor: Systagenix Wound Management (Industry)
Responsible Party: Sponsor
Other Study IDs: SBIR-001-B; Systagenix (Other: Systagenix)
Record Dates: First submitted 2013-06-11; First posted 2013-06-20 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Wounds
Keywords: Chronic wounds with different etiologies; Diabetic foot ulcers; venous leg ulcers; pressure sores; acute wounds
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer

STUDY DESIGN:
Biospecimen Retention: None Retained — Swabs will be tested on day on collection. Test is destructive. No swabs will be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment: No cohort as this study is not using a treatment or intervention only swabs are being collected.
  Interventions: Other: Swabs

INTERVENTIONS:
Other: Swabs — There is no intervention only swabs are being used to collect wound fluid samples

SUMMARY:
The objective of this study is to collect wound exudate (fluid) swab samples from Subjects who have wounds that show clinical signs of infection, as well as from Subjects who have wounds that do not show clinical signs of infection. Swab samples will be collected from acute and chronic wounds of different etiologies and these will be analysed for bacteria types and markers of infection.

ELIGIBILITY:
Inclusion Criteria:

* Subject has presented to participating study site with a wound(s) suspected to be infected, as determined by the Investigator and/ or study staff - defined as one that through clinical judgment has questionable infection status, and /or shows three or more of the NERDS or STONES signs of infection);
* Subject has presented to participating study site with a wound(s) suspected not to be infected, as determined by the Investigator and/ or study staff - defined as one that does not show three or more of the NERDS or STONES signs of infection.
* Subject is 18 years of age or older.
* Subject agrees to complete all aspects of the study and provides Informed Consent

Exclusion Criteria:

* Subject is less than 18 years of age.
* Target wound contains a malignancy
* Subject has hypersensitivity of the wound or painful wound surface which prevents touching/swabbing of the wound surface.
* Subject is confirmed to be positive for HIV or hepatitis.
* Subject is unable or unwilling to provide informed consent.
* Subjects deemed inappropriate for the study by the site's Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects (greater than 18 years old), presenting at participating clinical sites with wounds of different etiologies, who are willing to provide informed consent and who meet the inclusion / exclusion criteria, will be prospectively enrolled
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The determination of the protease levels in clinically infected and non infected chronic wounds from swabs by enzyme techniques. | 3 days
  Wound exudate (fluid) swab samples from different etiologies of wounds will be collected. Subjects who have wounds that do not show clinical signs of infection, as well as Subjects who have wounds that do show clinical signs of infection will be enrolled. a maximum of four (4) swab sample from Subjects from whom Informed Consent has been obtained. The swabs will be subjected to various tests methods that may include, but are not limited to, the following: 1) quantitative bacterial cultures (for aerobic and / or anaerobic bacteria), 2) "for research use only" testing on test formats currently in development by the sponsor (note: this data will not be used to support regulatory filings, such as CE marking or FDA submissions for U.S. market clearance), 3) molecular microbiology, and 4) protease analysis.

SECONDARY OUTCOMES:
to determine the bacteria present in infected and non infected wounds by microbiological techniques | 3 days
  The difference in the microbial flora will be determine by analysis of the swabs from infected and non infected wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Serena, MD, Principal Investigator — SerenaGroup, Inc.
Locations (1):
- St. John Wound Center, Tulsa, Oklahoma, United States